CLINICAL TRIAL: NCT06340789
Title: Functional Connectivity and Associated Neuropeptides Variations in Treatment Resistant Schizophrenia Patients: Treatment Efficacy of add-on Sodium Benzoate
Brief Title: Neurotransmitters in Treatment Resistant Schizophrenia Patients With add-on Sodium Benzoate
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-BR-110-49
Record Dates: First submitted 2021-11-03; First posted 2024-04-02 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-02

CONDITIONS: Symptom, Cognitive; Schizophrenia; Schizo Affective Disorder
Keywords: schizophrenia; sodium benzoate; cognition; treatment resistant schizophrenia
MeSH Terms: conditions — Neurobehavioral Manifestations; Schizophrenia; Psychotic Disorders; Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: The design and instrument are identical for two years. This add-on sodium benzoate randomized, double-blinded, placebo-controlled trial which is a two-arm, 6-week follow-up trial. The 90 patients will be 2:1 (SB: placebo) randomly assigned to 1. Treatment with sodium benzoate (A); or 2. placebo (P). The group of sodium benzoate treatment will be divided into two subgroups: 1. Responder (AR), and nonresponder (AN), as illustrated in Figure 4. The response criteria is defined the improvement of 20% total PANSS score after 6-week SB treatment. The participants with TRS will be enrolled in this trail from 3 hospitals(National Cheng Kung University Hospital, Tainan Hospital, Ministry of Health and Welfare, Chia-Yi branch, Taichung Veteran General Hospital).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment resistant schizophrenia patients with augmentation of sodium benzoate 2g/day (Active Comparator): with sodium benzoate 2g/day
  Interventions: Drug: Sodium Benzoate 2gram/day
- Treatment resistant schizophrenia patients with augmentation of placebo (Placebo Comparator): with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Benzoate 2gram/day — the add-on sodium benzoate with conventional pharmacological treatment
  Arms: Treatment resistant schizophrenia patients with augmentation of sodium benzoate 2g/day
Drug: Placebo — the add-on placebo with conventional pharmacological treatment
  Arms: Treatment resistant schizophrenia patients with augmentation of placebo

SUMMARY:
Although antipsychotic is effective for schizophrenia, however, still certain proportion of patients were not responsive to treatment. Treatment resistant schizophrenia (TRS) is accompanied by function decline and heavy burden. In recent decades, the biological mechanism of schizophrenia extended from dopamine theory to the role of glutamate system. This shift could be an alternative pathway to developing the treatment of TRS. Sodium benzoate (SB) could be an option as a glutamatergic agent for the patients with TRS. However, most evidence of SB is for treating patients with schizophrenia and other mental disorders but the evidence for treating patients with TRS is scarce. To predict the treatment response of SB will be an urgent topic in the future. Little is known about the precise medicine for treating patients with TRS. The present project will extend our pilot randomized clinical trial on SB for TRS. A total of 90 patients with TRS will be enrolled from three centers and will be assigned to 8 weeks of treatment with SB or placebo (2:1). A comprehensive battery of potential markers will be employed, including 1H- magnetic resonance spectroscopy (MRS), brain functional connectivity, genotyping, immune biomarkers, cognitive function, and clinical characteristics. The efficacy of SB on TRS will be confirmed in this project. Predictors for treatment response will be identified. Artificial intelligence algorithms will be used for probing the feasibility of precision medicine.

DETAILED DESCRIPTION:
The design and instrument are identical for two years. This add-on sodium benzoate randomized, double-blinded, placebo-controlled trial which is a two-arm, 6-week follow-up trial. The 90 patients will be 2:1 (SB: placebo) randomly assigned to 1. Treatment with sodium benzoate (A); or 2. placebo (P). The group of sodium benzoate treatment will be divided into two subgroups: 1. Responder (AR), and nonresponder (AN), as illustrated in Figure 4. The response criteria is defined the improvement of 20% total PANSS score after 6-week SB treatment. The participants with TRS will be enrolled in this trail from 3 hospitals(National Cheng Kung University Hospital, Tainan Hospital, Ministry of Health and Welfare, Chia-Yi branch, Taichung Veteran General Hospital).

ELIGIBILITY:
Inclusion Criteria:

1. Fulfil the DSM5 criteria for schizophrenia or schizoaffective disorder
2. Research criteria for treatment resistance: little or no symptomatic response to multiple (at least two) antipsychotic treatment of an adequate duration (at least 6 weeks) and adequate doses (equivalent to at least 600 milliequivalent (meq)/day of chlorpromazine)
3. 6 month period without remission (i.e. ≥4 item-score for the positive symptoms on PANSS scale , especially delusional thoughts, conceptual disorganisation, excitements, grandiosity, hallucinatory behaviour, excitement, persecution, and hostility)
4. The persistence of illness was defined as a score of ≥4 (moderately ill) on the severity of illness subscale of the Clinical Global Impression scale (CGI-S), and a lack of stable period of good social occupational function.

Exclusion Criteria:

1. Current or previous diagnosis of concurrent DSM-5 disorder due to active medical problems, known neurological disease, or a contraindication to MRI scanning
2. Current diagnosis of substance-related disorder
3. Any acute or chronic medical condition
4. History of head trauma or neurological diseases.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Brain imaging, functional MRI | 1hours
  All participants were scanned using a 1.5 Tesla GE scanner with eight channel head coils. 1H-MRS was performed to assess the concentrations of excitatory, glutamine, glutamate, glutamate complex (Glx), GABA and other neurometabolites. A three-dimensional T1-weighted inversion recovery magnetic resonance imaging (MRI) scan was performed in all participants, axial MRI three-dimensional brain volume, echo time (TE) = 2.9 ms, repetition time (TR) = 7.7, inversion time = 450 ms, flip angle = 12°, field of view =230 mm, matrix size = 256 × 256, and slice thickness = 1.0 mm

SECONDARY OUTCOMES:
Clinical psychiatric condition, Positive and Negative Symptoms Scale (PANSS) | 20 minutes
  The PANSS is a clinical tool used to measure symptom severity in patients with schizophrenia. It takes approximately 45 minutes to interview a patient with schizophrenia using the PANSS. The patient is rated from 1 to 7 on 30 different symptoms based on the interview, as well as descriptions of caregivers or hospital workers. There are seven positive symptoms, seven negative symptoms, and 16 general psychopathological traits.
Wechsler adult intelligence scales 4th edition (WAIS-IV) | 1 hours
  Specifically, for the cognitive function measurement, the WAIS-IV scale was used that comprises of five items: full-scale IQ (FSIQ), verbal comprehension index (VCI), perceptual reasoning index (PRI), WMI, and processing speed index (PSI), all of which are presented as different aspects of cognitive evaluation.
Continuous performance test third edition (CPT-3) | 20 minutes
  The CPT-3, is a computer assessment that evaluates attention-related deficits generally performed in ADHD. The test requires examinees to press the space bar when any letter appears, except for the letter "X." The entire test has 360 trials and takes approximately 14 minutes to administer. CPT-3 yields 10 Tscores: Omissions (OM), Variability (VAR), Commissions (COM), Perseveration (PER), Detectability (DET), Response Style (RS), Hit Reaction Time (HRT), HRT Block Change (BC), HRT Standard Deviation (HRT SD), and HRT Inter-Stimulus Interval (ISI) change, based on four different domains of attention: inattentiveness, impulsivity, sustained attention, and vigilance. The CPT-3 also includes an internal validity check which notifies the administrator that the administration is invalid if the examinee had too few hits on targets, an omission rate higher than 25%, or if there was a timing problem regarding administration.
Wisconsin card sorting test (WCST) | 20 minutes
  WCST Computer Version 4-Research Edition was used in this study, and patients were required to match response cards to four stimulus cards along one of three dimensions (colour, form, or number) on the basis of verbal feedback (correct or wrong) without providing any information about the dimensions. Once the subject sorted a series of 10 cards into one category, the subject was asked to sort the cards again by a different category. In the present study, 64 cards were used. All definitions of the indices have been described in the WCST manual.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Kuang Yang, Dr, Study Director — Psychiatry department, National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No